CLINICAL TRIAL: NCT03297047
Title: Randomized Controlled Trial Comparing Forearm and Upper Arm Combi Cast for Immobilization After Closed Reduced Distal Forearm Fractures in Children
Brief Title: Comparing Forearm and Upper Arm Combi Cast for Distal Forearm Fractures in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Principal Investigator, Georg Staubli, Dr. med., University Children's Hospital, Zurich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Forearm combi cast 2016
Record Dates: First submitted 2017-07-27; First posted 2017-09-29 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Salter-Harris Type I; Salter-Harris Type 2; Radius Fractures; Forearm Fracture
Keywords: cast, fracture, immobilization, displacement, child
MeSH Terms: conditions — Radius Fractures; Fractures, Bone

STUDY DESIGN:
Intervention Model Description: one Group with upper arm cast one Group with forearm cast
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- upper arm combi cast (Active Comparator): standardized treatment
  Interventions: Device: combi cast
- forearm combi cast (Experimental): Treatment with a forearm combi cast should be a sufficient immobilization
  Interventions: Device: combi cast

INTERVENTIONS:
Device: combi cast — upper arm or forearm combi cast

SUMMARY:
The standard treatment for children with closed reduction of displaced distal forearm fractures is an immobilization with an upper arm combicast. The hypothesis is that an forearm immobilization with combicast in children 4-16 years might be sufficient.

DETAILED DESCRIPTION:
Children with distal radial or forearm fractures needing closed reduction are eligible for this study. By drawing lots either an immobilization with an upper arm or forearm combicast will be performed. Regular controls after 5, 10, 28 days, 4 weeks and 7 weeks will be performed to check the rate of displacement, consolidation time, wearing comfort and movement of the elbow joint after taking off the cast.

ELIGIBILITY:
Inclusion Criteria:

* open growth Zone
* displaced metaphyseal radial or forearm fractures including Salter harris fracture 1 and 2 which require closed reduction
* written informed consent

Exclusion Criteria:

* intraarticular fractures
* open fractures
* unstable fractures

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2019-08-29 (Actual)

PRIMARY OUTCOMES:
secondary displacement of the fracture | Significant difference of secondary displaced fractures 28 days after closed reduction of fracture
  radiological evaluation

SECONDARY OUTCOMES:
Wearing comfort of the two different casts | 5, 10, 28 days, 4 weeks, 7 weeks after closed reduction of fracture
  help in daily life in hours
Mobilisation of elbow joint after cast removal | 4 weeks and 7 weeks after closed reduction of fracture
  Mobility of the elbow joint in degrees (flection and extension measurement)

CONTACTS AND LOCATIONS:
Overall Officials: Georg Staubli, Dr. med, Principal Investigator — Emergency department, University Children's Hospital Zurich
Locations (1):
- Children's Hospital, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Paneru SR, Rijal R, Shrestha BP, Nepal P, Khanal GP, Karn NK, Singh MP, Rai P. Randomized controlled trial comparing above- and below-elbow plaster casts for distal forearm fractures in children. J Child Orthop. 2010 Jun;4(3):233-7. doi: 10.1007/s11832-010-0250-1. Epub 2010 Mar 17. PMID 21629372
- [Background] Webb GR, Galpin RD, Armstrong DG. Comparison of short and long arm plaster casts for displaced fractures in the distal third of the forearm in children. J Bone Joint Surg Am. 2006 Jan;88(1):9-17. doi: 10.2106/JBJS.E.00131. PMID 16391244
- [Background] Boyer BA, Overton B, Schrader W, Riley P, Fleissner P. Position of immobilization for pediatric forearm fractures. J Pediatr Orthop. 2002 Mar-Apr;22(2):185-7. PMID 11856927
- [Background] Bhatia M, Housden PH. Re-displacement of paediatric forearm fractures: role of plaster moulding and padding. Injury. 2006 Mar;37(3):259-68. doi: 10.1016/j.injury.2005.10.002. Epub 2006 Jan 18. PMID 16414049
- [Background] Katz K, Weigl D, Becker T, Attias J, Bar-On E. Short-term after-effect of forearm cast removal in children. J Orthop Sci. 2011 May;16(3):283-5. doi: 10.1007/s00776-011-0054-2. Epub 2011 Mar 29. PMID 21590522
- [Derived] Seiler M, Heinz P, Callegari A, Dreher T, Staubli G, Aufdenblatten C. Short and long-arm fiberglass cast immobilization for displaced distal forearm fractures in children: a randomized controlled trial. Int Orthop. 2021 Mar;45(3):759-768. doi: 10.1007/s00264-020-04800-w. Epub 2020 Sep 17. PMID 32940750